CLINICAL TRIAL: NCT05370456
Title: The Adjunctive Use of Hyaluronic Acid for the Treatment of Multiple Adjacent Gingival Recessions With Coronally Advanced Flap Plus Xenogeneic Collagen Matrix: a Randomized Clinical Trial
Brief Title: Adjunctive Use of Hyaluronic Acid in Multiple Coronally Advanced Flap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XCM+HA_Turin
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Gingival Recession, Generalized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xenogenic collagen matrix (XCM) + Hyaluronic acid (HA) (Experimental): Multiple coronally advanced flap technique (mCAF) with the use of a XCM in combination with local application of a HA gel
  Interventions: Device: Local application of a HA gel for the treatment of MAGRs with mCAF technique and XCM
- Xenogenic collagen matrix (XCM) (Active Comparator): Multiple coronally advanced flap technique (mCAF) with the use of a XCM
  Interventions: Procedure: Treatment of MAGRs with mCAF technique and XCM

INTERVENTIONS:
Device: Local application of a HA gel for the treatment of MAGRs with mCAF technique and XCM — After local anaesthesia, mCAF technique with two releasing vertical incisions will be performed. XCM will be adapted on the root surfaces and positioned at the level of the cemento-enamel junction and HA gel will be applied.
  Arms: Xenogenic collagen matrix (XCM) + Hyaluronic acid (HA)
Procedure: Treatment of MAGRs with mCAF technique and XCM — After local anaesthesia, mCAF technique with two releasing vertical incisions will be performed. XCM will be adapted on the root surfaces and positioned at the level of the cemento-enamel junction.
  Arms: Xenogenic collagen matrix (XCM)

SUMMARY:
The primary aim of this study is to evaluate whether the effect of HA in combination with XCM for the treatment of MAGRs with a multiple coronally advanced flap technique (mCAF) achieves better results than the XCM with mCAF alone in terms of recession reduction (primary outcome) and other secondary root coverage outcomes (e.g. complete root coverage, mean root coverage). Moreover, this study aims to compare secondary clinical variables (e.g. keratinized tissue width (KTW) changes, probing pocket depth (PPD) changes, volumetric gain (VG), etc.), also with a digital approach, the patient-reported outcome measures (PROMs e.g. pain, swelling, bleeding) and lastly the expression of molecular mediators of tissue healing/regeneration. The hypothesis of this study is that at 6 months and 1 year follow-up the mCAF with XCM+HA is superior to the mCAF with only XCM in terms of recessions reduction and secondary clinical variables, including PROMs.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and able to sign informed consent
* At least 2 adjacent teeth with RT1 and/or RT2 gingival recessions without interproximal exposure of the CEJ (interdental gingival recession), at least one with a depth of ≥2mm with indication for root coverage treatment
* A minimum of 4 adjacent teeth (including the ones to be treated) in the region of interest
* Available to attend study related procedures (including follow-up visits)

Exclusion Criteria:

* Systemic diseases/medications which could influence the outcome of the therapy (e.g., uncontrolled diabetes mellitus);
* Current smokers (self-reported, any type of smoking), users of chewing tobacco, and drug/alcohol abusers;
* Pregnant or nursing women;
* History of previous periodontal surgery (mucogingival or other) on the teeth to be included;
* Furcation involvement in the teeth to be included;
* Presence of severe tooth malposition, rotation or clinically significant extrusion in the teeth to be treated;
* Presence of fixed or removable prosthesis in the area to be treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-09-10 (Estimated); Study Completion 2024-09-10 (Estimated)

PRIMARY OUTCOMES:
Mean Recession Reduction (RecRed) | 6 months; 1 year
  Mean changes in mm in recession depth between baseline and 1-year

SECONDARY OUTCOMES:
Complete Root Coverage (CRC) | 6 months; 1 year
  Percentage of sites with complete root coverage after 1-year
Mean Root Coverage (MRC) | 6 months; 1 year
  Percentage of mean root coverage after 1-year
Keratinised tissue height (KTH) changes | 6 months; 1 year
  Linear changes in mm from the gingival margin to the mucogingival junction between baseline and 1-year
Post-operative morbidity (pain, swelling, discomfort) | 14 days
  Assessment of patient's pain, swelling and discomfort at 14 days after the procedure using visual analogue scale (VAS) ranging from 0 (no pain, swelling or discomfort) to 10 (maximum pain, swelling or discomfort) with a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: Undecided